CLINICAL TRIAL: NCT00700375
Title: Prevention of Contrast-Induced Nephropathy With Sodium Bicarbonate Bolus Injection in Patients Undergoing an Emergent Coronary Procedure
Brief Title: Prevention of Contrast-Induced Nephropathy With Sodium Bicarbonate Bolus Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Osaka General Medical Center (Other)
Responsible Party: Hiromichi Ueda, Osaka General Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SBECP
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Results first posted 2010-07-09 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-03

CONDITIONS: Emergent Coronary Procedure
Keywords: Patients undergoing an emergent coronary procedure
MeSH Terms: interventions — Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium bicarbonate (Experimental)
  Interventions: Drug: Sodium bicarbonate
- Sodium chloride (Experimental)
  Interventions: Drug: Sodium Chloride

INTERVENTIONS:
Drug: Sodium bicarbonate — 8.4%sodium bicarbonate 0.5ml/kg bolus injection before procedure and hydration with 154mEq/l sodium bicarbonate 1ml/kg/Hr for 6 hours after the procedure
  Arms: Sodium bicarbonate
Drug: Sodium Chloride — 8.4%sodium bicarbonate 0.5ml/kg bolus injection before procedure and hydration with 154mEq/l sodium bicarbonate 1ml/kg/Hr for 6 hours after the procedure
  Arms: Sodium chloride

SUMMARY:
This study is to investigate the effect of Sodium Bicarbonate bolus injection in patients undergoing an emergent coronary procedure for prevention of contrast-induced nephropathy.

DETAILED DESCRIPTION:
This study is to investigate the effect of Sodium Bicarbonate bolus injection in patients undergoing an emergent coronary procedure for prevention of contrast-induced nephropathy.The End point is development of contrast-induced nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an emergent coronary procedure(within 60 minutes from admission)

Exclusion Criteria:

* On dialysis
* Pregnancy
* Past use of bicarbonate or N-Acetyl-Cystein in 48hr
* Past exposure to contrast media in 48hr
* Circulatory insufficiency with lactic acidosis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takahisa Yamada, directorate, Study Chair — OsakaGeneralMedicalCenter
Locations (1):
- Osaka General Medical Center, Osaka, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Sodium Bicarbonate Group: Randomly assigned to the sodium bicarbonate group or the sodium chloride group in a single-blinded fashion. This group received an intravenous bolus injection of sodium bicarbonate with a dose of 0.5ml/kg as soon as possible before the administration of contrast medium. Afterward, the both groups were followed by an intravenous infusion of 1 ml/kg/hour sodium bicarbonate during and for 6 hours after the procedure.Nonionic, low-osmolality nonionic contrast media were used in all procedure and the volumes were left to the discretion of the operator. Emergent coronary procedures were almost performed by femoral approach. The decision to use an intra-aortic balloon pump, inotropic drugs, beta blockers, angiotensin-convertiong enzyme inhibitors, angiotensin receptor blockers or diuretics was based on international guidelines and left to the discretion of the attending physician.
- Sodium Chloride Group: This group received an intravenous bolus injection of sodium chloride with a dose of 0.5ml/kg as soon as possible before the administration of contrast medium. Afterward, the both groups were followed by an intravenous infusion of 1 ml/kg/hour sodium bicarbonate during and for 6 hours after the procedure.Nonionic, low-osmolality nonionic contrast media were used in all procedure and the volumes were left to the discretion of the operator. Emergent coronary procedures were almost performed by femoral approach. The decision to use an intra-aortic balloon pump, inotropic drugs, beta blockers, angiotensin-convertiong enzyme inhibitors, angiotensin receptor blockers or diuretics was based on international guidelines and left to the discretion of the attending physician.
Period: Overall Study
Arm/Group | Sodium Bicarbonate Group | Sodium Chloride Group
Started | 30 | 29
2 Days After Creatinine Mesurement | 30 | 29
Completed | 30 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Bicarbonate Group | Sodium Chloride Group | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 11
  >=65 years | 26 | 22 | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 76 (9.3) | 75 (10.3) | 75 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 23 | 23 | 46
Region of Enrollment [Number; unit: participants]
  Japan | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Contrast-induced Nephropathy
Description: The primary endpoint was the occurrence of contrast-induced nephropathy, defined as an increase >0.5 mg/dl or >25% in serum Cr concentration within 2 days of the procedure compared to the baseline level.
Time Frame: after procedure and 1,2-3day after procedure
Measure: Number; unit: participants
Arm/Group | Sodium Bicarbonate Group | Sodium Chloride Group
Number analyzed (Participants) | 30 | 29
participants | 1 | 8

ADVERSE EVENTS:
Time Frame: 1 month
Description: lethal arrhythmia and death
Arm/Group | Sodium Bicarbonate Group | Sodium Chloride Group
Serious Adverse Events (participants affected / at risk) | 2/30 | 3/29
Other Adverse Events (participants affected / at risk) | 0/30 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Bicarbonate Group (N=30) | Sodium Chloride Group (N=29)
lethal arrhythmia and death (Cardiac disorders) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
Single center trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes